CLINICAL TRIAL: NCT01667952
Title: Prospective Ascertainment for Late Effects Among Survivors of Cancer, Tumor, or a Related Illness
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-143
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pediatric or Young Adult Cancer Survivors
Keywords: Family History Questionnaire (FHQ); Blood sample; Salvia sample; 12-145
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva or blood samples will be collected in the clinic at the time of a routine visit.

GROUPS / COHORTS (1):
- Cancer Survivors: The purpose of this study is to establish a registry of survivors of cancer, tumors,or a related illness. The registry will include detailed family history and germline DNA. Ultimately, we hope to improve our understanding of genetic susceptibility to secondary malignant neoplasms and other late effects among survivors of cancer, tumors, or a related illness.
  Interventions: Genetic: Family History Questionnaire (FHQ); Genetic: Salvia sample; Other: Blood sample

INTERVENTIONS:
Genetic: Family History Questionnaire (FHQ) — Consented subjects will be given the Family History Questionnaire (FHQ) to complete either in clinic or at home. Subjects who chose to complete the FHQ at home will be given a stamped envelope with a label. For participants who are children and cannot fill out the questionnaire on their own, the clinic RSA will instruct the parent, guardian, or legally authorized representative (LAR) present to fill out the questionnaire, reminding them that the "You" in the questionnaire refers to their child.
Genetic: Salvia sample — The saliva samples will be collected in Oragene DNA Self-Collection Kits or a similar product. Patients will be instructed to donate about 2ml of saliva into a vial, which contains 2ml of product. Oragene or similar solution.
Other: Blood sample — Subjects will be offered the option of a blood collection instead of saliva. For adult subjects who opt for blood collection, two tubes of blood (approximately 20cc) will be drawn from the utilizing a sterile technique. For subjects under the age of 18 who opt for blood collection, approximately 3-5cc of blood will be collected utilizing a sterile technique.

SUMMARY:
The purpose of this study is to establish a registry of survivors of cancer, tumor, or a related illness.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* A personal history of cancer tumor, or a related illness
* Followed in the the Adult Long Term Follow Up Program, Pediatric Long Term Follow Up Program, or Lymphoma Service at MSKCC

Exclusion Criteria:

* Evidence of active progression of disease or recurrence
* Neurocognitive deficits that impair ability to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Adult Long-Term Follow-Up Program, the Pediatric Long Term Follow-up Program, or Lymphoma Service will be recruited at a routine visit to MSKCC.
Sampling Method: Non-Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2012-08; Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
establish a registry of DNA | 4 years
  For the purpose of facilitating future genetic laboratory investigations of late effects among of survivors of cancer, tumors, or a related illness. Patients in the ALTFU Program are followed for secondary malignant neoplasms and other adverse outcomes (so-called "late effects") including cardiomyopathy, pulmonary fibrosis, cardiac valvular pathology, osteoporosis, and others. The following data will be ascertained from each study participant: (1) family history information will be ascertained using the Family History Questionnaire (Appendix A); and (2) saliva or blood samples for genetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friedman, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/